CLINICAL TRIAL: NCT04726683
Title: Trigger Point Dry Needling vs Injection in Patients With Temporomandibular Disorders: a Randomized Placebo-controlled Trial
Brief Title: Dry Needling vs Injection in Patients With Temporomandibular Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Josue Fernandez Carnero (Other)
Responsible Party: Sponsor-Investigator, Josue Fernandez Carnero, Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC-09/2020
Record Dates: First submitted 2020-11-13; First posted 2021-01-27 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Temporomandibular Disorders
Keywords: dry needling; Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Dry Needling; Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dry needling (Experimental): Trigger point dry needling on an active myofascial trigger point of the masseter muscle.
  Interventions: Procedure: Dry needling and placebo injection
- Injection (Experimental): Trigger point injection of lidocaine on an active myofascial trigger point of the masseter muscle.
  Interventions: Procedure: Injection and placebo dry needling
- Placebo (Placebo Comparator): Combines sham dry needling + sham injection.
  Interventions: Procedure: Placebo dry needling and placebo injection
- Dry needling + Injection (Active Comparator): Combines experimental dry needling and injection
  Interventions: Procedure: Dry needling and injection

INTERVENTIONS:
Procedure: Dry needling and placebo injection — Dry Needling is applied with a filiform needle to penetrate the skin and stimulate the underlying myofascial trigger point of the masseter muscle. Dry needling is combined with placebo injection, in which the tip of a beveled needle is cut and the process of injection is simulated without penetrating the skin.
  Arms: Dry needling
Procedure: Injection and placebo dry needling — Lidocaine injection applied in the myofascial trigger point of the masseter muscle. Lidocaine injection is combined with placebo dry needling, in which the tip of a filiform needle is cut and the dry needling technique simulated without penetrating the skin
  Arms: Injection
Procedure: Dry needling and injection — Dry Needling is applied with a filiform needle to penetrate the skin and stimulate the underlying myofascial trigger point of the masseter muscle. Dry needling is combined with lidocaine injection applied in the myofascial trigger point of the masseter muscle.
  Arms: Dry needling + Injection
Procedure: Placebo dry needling and placebo injection — Placebo dry needling, in which the tip of a filiform needle is cut and the dry needling technique simulated without penetrating the skin. Placebo dry needling is combined with placebo injection, in which the tip of a beveled needle is cut and the process of injection is simulated without penetrating the skin
  Arms: Placebo

SUMMARY:
The main objective is to compare the effectiveness of dry needling in improving pain and disability versus placebo, and versus infiltration, in patients with myofascial temporomandibular dysfunction in the short, medium and long term.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 60 years.
2. Pain of more than 6 weeks of evolution in the craniofacial region.
3. TMD with origin in the masticatory musculature according to the "DC-TMD" criteria.

Exclusion Criteria:

1. Previous injection or dry needling intervention (3 months) on the masseter muscle.
2. Arthrogenous TMD.
3. History of trauma, infection in the temporomandibular joint in the last 6 months.
4. Coagulation disorders.
5. Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain perception (Change is being assessed) | At baseline, 24h post treatment, at one month, at six months and at twelve months
  Self reported Visual Analog Scale. Minimum value is 0 (best); Maximun value is 10 (worst).

SECONDARY OUTCOMES:
Believability of placebo | At one week, at two weeks, at three weeks, at for weeks
  Patients beliefs about group allocation: A scale of cale of four options (Experimental Dry needling / Experimental Injection / Placebo Comparator / Active Comparator) in which patients had to indicate which intervention they believe they have received during the treatment sessions.
Disability | At baseline, 24h post treatment, at one month, at six months and at twelve months
  Self-reported disability questionnaire: Craniofacial Pain and Disability Inventory (CF-PDI).
  The CF-PDI contains 21 items divided into 2 subscales according to their content and exploratory factor analysis: "pain and disability" and "jaw functional status."
Pressure pain threshold (Change is being assessed) | At baseline, 24h post treatment, at one month, at six months and at twelve months
  Digital algometer measure of the pressure pain threshold on the masseter muscle
Conditioned pain modulation | At baseline, 24h post treatment, at one month, at six months and at twelve months
  Pressure pain thresholds measure on the distal phalanx of the thumb before and during the application of a noxious stimulus ( Ischemic pain)
Temporal summation (TS) | At baseline, 24h post treatment, at one month, at six months and at twelve months
  Initially, a needlle stimulus is measured locally and distally. Then, the TS is triggered by 10 consecutive pressures on the PPT at the pressure determined at each location. For each pulse, the pressure was gradually increased at a rate of 2 kg/s at the determined PPT and held for 1 s before being released (with an interval of one second between each stimulus).
Beck Depression Inventory (BDI) | At baseline, 24h post treatment, at one month, at six months and at twelve months
  The level of depressive symptomatology was measured by the Spanish version of the Beck Depression Inventory (BDI-II); a 21-item self-report rating scale that assesses affective, cognitive and somatic symptoms of depression. Each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms.
Anxiety (STAI questionnaire) | At baseline, 24h post treatment, at one month, at six months and at twelve months
  The state-trait anxiety inventory (STAI) is a questionnaire that measures trait anxiety (a personality factor that predisposes the patient to suffer from anxiety) and the state of anxiety (environmental factors that protect or generate anxiety). Each of the two sub-scales (trait anxiety and state anxiety) consists of 20 items, ranging from 0 (nothing) to 3 (a lot).
Kinesiophobia (TAMPA scale) | At baseline, 24h post treatment, at one month, at six months and at twelve months
  Tampa Scale for Kinesiophobia. To assess the fear of movement and pain-related fear. The 11 items are scored 1-4, with total scores ranging from 11 to 44. The addition of all the points obtained from each of the items results in the level of kinesiophobia, with higher scores indicating greater perceived kinesiophobia
Fair avoidance beliefs (FAB questionnaire) | At baseline, 24h post treatment, at one month, at six months and at twelve months
  Fear-avoidance Beliefs Questionnaire . The instrument consists of two subscales, a four-item physical activity subscale, and a seven-item work subscale. Each item is scored from 0 to 6 and summed to produce the subscale score. Possible scores range from 0-28 to 0-42, with higher scores indicating greater fear avoidance beliefs.
Pain catastrophizing (PCS) | At baseline, 24h post treatment, at one month, at six months and at twelve months
  Pain catastrophizing Scale (PCS). This tool is a 13-item questionnaire designed to measure the three components of pain-related catastrophizing: rumination, magnification, and helplessness, resulting in a unique score. Each item is responded to on a 5-point scale (0 not at all, 4 all the time) relating the degree to which the individual experiences a thought or feeling of a painful situation.
Expectation of improvement | Baseline, at one week, at two weeks, at three weeks, at for weeks
  Patients´ expectations of pain improvement after the intervention. Patients report their estimated pain perception after the treatment by completing a Self reported Visual Analog Scale. Minimum value is 0 (best); Maximun value is 10 (worst).
Central sensitization inventory | At baseline, 24h post treatment, at one month, at six months and at twelve months
  It serves to identify the symptoms related to central sensitization. It consists of 25 items that are scored from 0: never to 4: always reaching a maximum score of 100. Results are interpreted as follows: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100.
Mandibular Dynamic | At baseline, 24h post treatment, at one month, at six months and at twelve months
  Interincisal distance measured in cm.
Neuropathic pain | At baseline, 24h post treatment, at one month, at six months and at twelve months
  The presence of neuropathic pain will be assessed using the DN4 questionnaire validated in Spanish. This clinician-administered questionnaire consists of 10 questions. Seven of them are related to the quality of pain and are based on the patient interview, and the remaining three are based on clinical examination according to the presence or absence of hypoesthesia and tactile allodynia to pressure and touch.
Pain body map | At baseline, 24h post treatment, at one month, at six months and at twelve months
  The patient will be asked to paint the areas where he/she presents pain. This map consists of a representation of a person drawn in an anterior, posterior and two lateral planes. The drawing is in a grid of 10mm x 10mm, 16mm x 16 mm cells, up to a maximum of 256 cells.
EQ-5D | At baseline, 24h post treatment, at one month, at six months and at twelve months
  . It consists of two parts: the descriptive EQ-5D system and the VAS. It is a generic and standardized questionnaire, self-administered, simple to answer and with low cognitive load.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Universitaria de la Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain